CLINICAL TRIAL: NCT01517373
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled, Dose-ranging, Parallel Group Study To Evaluate Safety And Efficacy Of Pf-04937319 And Glimepiride In Adult Patients With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Study To Understand Efficacy And Safety Of Investigational Agent (PF-04937319) Compared To Approved Agent (Glimepiride) In Patients With Diabetes On Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1621002; 2011-005206-30 (EudraCT Number)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: T2DM; PF-04937319; Phase 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo to match PF-04937319 and glimepiride
  Interventions: Drug: Placebo
- PF-04937319 10 mg (Experimental)
  Interventions: Drug: PF-04937319 10 mg
- PF-04937319 50 mg (Experimental)
  Interventions: Drug: PF-04937319 50 mg
- PF-04937319 100 mg (Experimental)
  Interventions: Drug: PF-04937319 100 mg
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Placebo — Combination of tablets and capsules, a total of 3 pills/dose, administered once daily for 84-days
  Arms: Placebo
Drug: PF-04937319 10 mg — Combination of tablets and capsules, dose of 10 mg, a total of 3 pills/dose, administered once daily for 84-days
  Arms: PF-04937319 10 mg
Drug: PF-04937319 50 mg — Combination of tablets and capsules, dose of 50 mg, a total of 3 pills/dose, administered once daily for 84-days
  Arms: PF-04937319 50 mg
Drug: PF-04937319 100 mg — Combination of tablets and capsules, dose of 100 mg, a total of 3 pills/dose, administered once daily for 84-days
  Arms: PF-04937319 100 mg
Drug: Glimepiride — Combination of tablets and capsules, dose of up to 6 mg, a total of 3 pills/dose, administered once daily for 84-days
  Arms: Glimepiride

SUMMARY:
This is a study to understand efficacy and safety of investigational agent (PF-04937319) compared to approved agent (glimepiride) in patients with diabetes on metformin

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs, male and females, with T2DM, on metformin alone or in combination with 1 other oral agent

Exclusion Criteria:

* Subjects with recent cardiovascular events, those with evidence of diabetic complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (23):
  - Sierra Clinical Research, Roseville, California
  - California Research Foundation, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Meridien Research, Bradenton, Florida
  - South Broward Research, LLC, Pembroke Pines, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Center of Cape Cod, Inc., Hyannis, Massachusetts
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Diagnostic Center, Chattanooga, Tennessee
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Bristol Clinical Research, LLC, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - Aurora Advanced Healthcare, Inc., Milwaukee, Wisconsin
- Bulgaria (6):
  - MBAL Yulia Vrevska - Byala, Otdelenie po vatreshni bolesti, Byala
  - MBAL - Ruse AD, Vtoro otdelenie po vatreshni bolesti, Rousse
  - DKTs Akta Medika, Kabinet po endokrinologia, Sevlievo
  - UMBAL Aleksandrovska, Klinika po endokrinologia i bolesti na obmyanata, Sofia
  - VMA - MBAL - Sofia, Klinika po endokrinologia i bolesti na obmyanata, Sofia
  - UMBAL Stara Zagora, Klinika po endokrinologia i bolesti na obmyanata, Stara Zagora
- Canada (9):
  - Glover Medical Clinic, Langley, British Columbia
  - Ocean West Research Clinic Inc., Surrey, British Columbia
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Aggarwal and Associates Limited, Brampton, Ontario
  - DCTM CLinical Trials Group Ltd., Strathroy, Ontario
  - Manna Research, Toronto, Ontario
  - Alpha Recherche Clinique, Québec, Quebec
  - Pro-Recherche, Saint Romuald, Quebec
  - Centre de cardiologie et de Recherche Clinique Pierre-Le Gardeur, Terrebonne, Quebec
- Hungary (4):
  - Dr. Kenessey Albert Korhaz-Rendelointezet/Belgyogyaszat, Balassagyarmat
  - Synexus Magyarorszag Kft., Budapest
  - Semmelweis Egyetem/I. sz. Belgyogyaszati Klinika, Budapest
  - Fejer Megyei Szent Gyorgy Korhaz/II. Belgyogyaszati Osztaly, Székesfehérvár
- India (3):
  - BGS Global Hospital, Bangalore, Karnataka
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Diabetes Unit, K.E.M. Hospital Research Centre, Pune, Maharashtra
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Interna A Diabetologicka Ambulancia, Moldava nad Bodvou
  - FUNKYSTUFF, s.r.o., Nové Zámky
  - MEDIAB, s.r.o., Pezinok
  - MEDIVASA, s.r.o., Žilina
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

REFERENCES:
- [Derived] Amin NB, Aggarwal N, Pall D, Paragh G, Denney WS, Le V, Riggs M, Calle RA. Two dose-ranging studies with PF-04937319, a systemic partial activator of glucokinase, as add-on therapy to metformin in adults with type 2 diabetes. Diabetes Obes Metab. 2015 Aug;17(8):751-9. doi: 10.1111/dom.12474. Epub 2015 May 11. PMID 25885172
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621002&StudyName=Study%20To%20Understand%20Efficacy%20And%20Safety%20Of%20Investigational%20Agent%20%28PF-04937319%29%20Compared%20To%20Approved%20Agent%20%28Glimepiride%29%20In%20Patients%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 628 participants were consented. Of these, 361 participants transitioned to the run-in period and received sponsor provided background therapy of Metformin. Participants completed the run-in period were then randomized to receive either placebo, PF-04937319 (10, 50 or 100 milligram [mg]) or Glimepiride in treatment period.
Groups:
- Metformin 500 mg: Metformin 500 milligram (mg) immediate release tablet used as standardized, pre-specified background therapy in all participants initiated at the run-in visit and continued till follow-up visit.
- Placebo: Placebo matched to PF-04937319 tablet and placebo matched to glimepiride oral capsule once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 10 mg: PF-04937319 10 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 50 mg: PF-04937319 50 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 100 mg: PF-04937319 100 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- Glimepiride: Glimepiride capsule at a starting dose of 2 milligram per day (mg/day) up to a maximum dose of 6 mg/day along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
Period: Run-in Period
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Started | 361 | 0 | 0 | 0 | 0 | 0
Completed | 304 | 0 | 0 | 0 | 0 | 0
Not Completed | 57 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet eligibility criteria | 34 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Started | 0 | 61 | 60 | 61 | 61 | 61
Completed | 0 | 57 | 54 | 54 | 55 | 54
Not Completed | 0 | 4 | 6 | 7 | 6 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 2 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 3 | 2 | 0
Not completed — Medication error without AEs | 0 | 0 | 2 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride | Total
Number analyzed (Participants) | 61 | 60 | 61 | 61 | 61 | 304
Age, Customized [Number; unit: participants]
  >=18 to =<44 years | 8 | 4 | 8 | 11 | 7 | 38
  >=45 to =<64 years | 45 | 48 | 40 | 35 | 48 | 216
  >64 years | 8 | 8 | 13 | 15 | 6 | 50
Gender [Count of Participants; unit: Participants]
  Female | 27 | 26 | 24 | 32 | 22 | 131
  Male | 34 | 34 | 37 | 29 | 39 | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1C) at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average glycemic control over prolonged periods of time. The normal range for the HbA1c test, was identified as less than 6.5 percent by the study-specific central laboratory used. Change from baseline in percentage of HbA1C was reported.
Time Frame: Baseline (Day 1), Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure and 'n' signifies participants evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 59 | 57 | 55 | 60 | 60
percentage of hemoglobin
  Baseline (n=59, 57, 55, 60, 60) | 7.90 (0.988) | 7.97 (0.886) | 7.91 (0.987) | 7.88 (0.969) | 8.12 (0.884)
  Change at Week 12 (n=56, 53, 53, 54, 54) | -0.13 (0.789) | -0.18 (0.804) | -0.45 (0.733) | -0.64 (0.797) | -1.01 (0.709)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 10 mg; Treatment difference and 80 percent (%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment,duration of type 2 diabetes mellitus (T2DM),time and treatment-by-time interaction as fixed effects,baseline as the covariate,time was repeated for participant. Null hypothesis stated there was no difference between PF 04937319 and placebo, alternative hypothesis stated PF 04937319 was superior to placebo; Test type: Superiority or Other; p = 0.4468, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; Least Squares (LS) Mean Difference = -0.02, 80% CI 2-sided [-0.21 to 0.17], Standard Error of Mean 0.145
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 50 mg; Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant. Null hypothesis stated there was no difference between PF 04937319 and placebo, alternative hypothesis stated PF 04937319 was superior to placebo; Test type: Superiority or Other; p = 0.0218, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; LS Mean Difference = -0.30, 80% CI 2-sided [-0.48 to -0.11], Standard Error of Mean 0.146
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0006, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; LS Mean Difference = -0.47, 80% CI 2-sided [-0.65 to -0.28], Standard Error of Mean 0.144
Statistical Analysis 4: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; LS Mean Difference = -0.83, 80% CI 2-sided [-1.02 to -0.65], Standard Error of Mean 0.144

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1C) at Week 2, 4, 6 and 8
Description: as for outcome 1
Time Frame: Baseline (Day 1), Week 2, 4, 6, 8
Population: FAS: All randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was summarized for this measure and 'n' signifies participants who were evaluable at given time points for each group. Data for Week 2 had not been reported because as per protocol it was not intended to be collected.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 58 | 57 | 55 | 58 | 60
percentage of hemoglobin
  Week 4 (n=58, 57, 55, 58, 60) | -0.08 (0.590) | -0.07 (0.422) | -0.22 (0.431) | -0.32 (0.532) | -0.54 (0.379)
  Week 6 (n=57, 55, 55, 58, 55) | -0.14 (0.676) | -0.14 (0.545) | -0.22 (0.494) | -0.51 (0.479) | -0.78 (0.500)
  Week 8 (n=58, 55, 53, 57, 55) | -0.19 (0.756) | -0.17 (0.628) | -0.38 (0.575) | -0.59 (0.571) | -0.89 (0.582)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 10 mg; Week 4: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.6112, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = 0.02, 80% CI 2-sided [-0.09 to 0.14], Standard Error of Mean 0.087
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0550, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.14, 80% CI 2-sided [-0.25 to -0.03], Standard Error of Mean 0.088
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 100 mg; Week 4: Treatment difference and 80%CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.0032, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.24, 80% CI 2-sided [-0.35 to -0.13], Standard Error of Mean 0.086
Statistical Analysis 4: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.44, 80% CI 2-sided [-0.55 to -0.33], Standard Error of Mean 0.086
Statistical Analysis 5: Comparison: Placebo vs PF-04937319 10 mg; Week 6: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.6146, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = 0.03, 80% CI 2-sided [-0.10 to 0.16], Standard Error of Mean 0.101
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.2606, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.07, 80% CI 2-sided [-0.19 to 0.06], Standard Error of Mean 0.101
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0006, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.32, 80% CI 2-sided [-0.45 to -0.20], Standard Error of Mean 0.099
Statistical Analysis 8: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.57, 80% CI 2-sided [-0.70 to -0.44], Standard Error of Mean 0.100
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 10 mg; Week 8: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.6618, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = 0.05, 80% CI 2-sided [-0.10 to 0.20], Standard Error of Mean 0.118
Statistical Analysis 10: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0878, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.16, 80% CI 2-sided [-0.31 to -0.01], Standard Error of Mean 0.119
Statistical Analysis 11: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0022, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.34, 80% CI 2-sided [-0.49 to -0.19], Standard Error of Mean 0.117
Statistical Analysis 12: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -0.66, 80% CI 2-sided [-0.81 to -0.51], Standard Error of Mean 0.117

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 2, 4, 6, 8 and 12
Time Frame: Baseline (Day 1), Week 2, 4, 6, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure and 'n' signifies participants evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 60 | 59 | 60 | 61 | 61
milligram per deciliter (mg/dL)
  Baseline (n=60, 59, 60, 61, 61) | 161.3 (30.74) | 168.7 (43.01) | 174.7 (36.43) | 160.4 (37.03) | 163.7 (35.99)
  Change at Week 2 (n=60, 59, 60, 61, 59) | 3.1 (23.89) | -2.0 (46.24) | -7.9 (29.29) | -10.5 (20.83) | -19.9 (25.68)
  Change at Week 4 (n=59, 58, 56, 59, 60) | -0.5 (27.66) | -8.4 (41.99) | -7.7 (27.49) | -11.4 (22.84) | -26.2 (31.00)
  Change at Week 6 (n=58, 56, 56, 59, 57) | -2.6 (31.40) | -6.9 (41.80) | -7.2 (24.63) | -10.4 (28.48) | -23.4 (35.01)
  Change at Week 8 (n=59, 56, 54, 58, 57) | 0.9 (29.70) | -7.0 (43.93) | -13.0 (27.48) | -13.0 (23.07) | -26.9 (32.08)
  Change at Week 12 (n=57, 54, 54, 55, 55) | 3.4 (31.29) | -6.2 (45.22) | -9.9 (37.09) | -10.3 (34.69) | -22.5 (30.86)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 10 mg; Week 2: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.3446, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -2.09, 80% CI 2-sided [-8.80 to 4.62], Standard Error of Mean 5.222
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1204, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -6.12, 80% CI 2-sided [-12.81 to 0.57], Standard Error of Mean 5.210
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0041, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -13.74, 80% CI 2-sided [-20.37 to -7.10], Standard Error of Mean 5.166
Statistical Analysis 4: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -21.34, 80% CI 2-sided [-28.01 to -14.67], Standard Error of Mean 5.192
Statistical Analysis 5: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1616, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -5.14, 80% CI 2-sided [-11.80 to 1.53], Standard Error of Mean 5.191
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1974, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -4.45, 80% CI 2-sided [-11.15 to 2.26], Standard Error of Mean 5.219
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0122, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -11.62, 80% CI 2-sided [-18.22 to -5.02], Standard Error of Mean 5.140
Statistical Analysis 8: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -24.79, 80% CI 2-sided [-31.37 to -18.20], Standard Error of Mean 5.129
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3645, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -1.97, 80% CI 2-sided [-9.26 to 5.32], Standard Error of Mean 5.674
Statistical Analysis 10: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3672, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -1.93, 80% CI 2-sided [-9.22 to 5.36], Standard Error of Mean 5.676
Statistical Analysis 11: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0906, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -7.50, 80% CI 2-sided [-14.69 to -0.31], Standard Error of Mean 5.598
Statistical Analysis 12: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0003, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -19.69, 80% CI 2-sided [-26.91 to -12.46], Standard Error of Mean 5.624
Statistical Analysis 13: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.1748, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -5.18, 80% CI 2-sided [-12.29 to 1.93], Standard Error of Mean 5.534
Statistical Analysis 14: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0297, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -10.54, 80% CI 2-sided [-17.69 to -3.38], Standard Error of Mean 5.566
Statistical Analysis 15: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0118, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -12.44, 80% CI 2-sided [-19.47 to -5.41], Standard Error of Mean 5.469
Statistical Analysis 16: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -27.00, 80% CI 2-sided [-34.04 to -19.96], Standard Error of Mean 5.480
Statistical Analysis 17: Comparison: Placebo vs PF-04937319 10 mg; Week 12: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.1012, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -8.03, 80% CI 2-sided [-16.10 to 0.04], Standard Error of Mean 6.281
Statistical Analysis 18: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.0409, t-test, 1 sided; LS Mean Difference = -10.99, 80% CI 2-sided [-19.07 to -2.91], Standard Error of Mean 6.287
Statistical Analysis 19: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.0089, t-test, 1 sided; LS Mean Difference = -14.87, 80% CI 2-sided [-22.88 to -6.86], Standard Error of Mean 6.232
Statistical Analysis 20: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — P-value was 1-sided; LS Mean Difference = -25.93, 80% CI 2-sided [-33.93 to -17.92], Standard Error of Mean 6.233

4. Secondary Outcome: Percentage of Participants Achieving Less Than 6.5 Percent and Less Than 7 Percent Glycosylated Hemoglobin (HbA1c) Levels at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average glycemic control over prolonged periods of time. The normal range for the HbA1c test, was identified as less than 6.5 percent by the study-specific central laboratory used and data are presented in categories of less than 6.5 percent and less than 7 percent.
Time Frame: Week 12
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 57 | 54 | 54 | 55 | 55
percentage of participants
  Less Than 6.5 Percent | 7.0 | 13 | 18.5 | 27.3 | 18.2
  Less Than 7 Percent | 26.3 | 31.5 | 27.8 | 52.7 | 45.5

5. Secondary Outcome: Number of Participants With Increase From Baseline Electrocardiogram (ECG) Data
Description: Participants who met the criteria for increase from baseline in ECG data were reported. Criteria for increase from baseline data: PR interval (percent change of greater than or equal to [>=] 25/50% [if baseline value was >200 then percent change of >25% counts; if baseline value was <=200 then percent change of >50% counts]); QRS complex (percent change of >=50%); QT Fridericia's correction (QTcF) interval (change of >= 30 to <60 millisecond [msec], and change of >=60 msec).
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. N(number of participants analyzed)= participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 60 | 59 | 59 | 61 | 61
participants
  PR interval: Percent change of >=25/50% | 0 | 0 | 1 | 0 | 0
  QRS interval: Percent change of >=50% | 0 | 1 | 1 | 2 | 1
  QTcF interval: Change of >=30 to <60 msec | 6 | 5 | 8 | 6 | 4
  QTcF interval: Change of >=60 msec | 2 | 2 | 2 | 2 | 1

6. Secondary Outcome: Number of Participants With Increase/Decrease From Baseline Vital Signs Data
Description: Participants who met the criteria for increase or decrease in vital signs data were reported. Criteria for increase or decrease from baseline vital signs data: sitting systolic blood pressure (BP) of >=30 millimeter of mercury (mmHg); sitting diastolic BP of >=20 mmHg and pulse rate was based on investigator's discretion.
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 60 | 60 | 60 | 61 | 61
participants
  Increase in systolic BP (>=30 mmHg) | 2 | 1 | 3 | 3 | 5
  Increase in diastolic BP (>=20 mmHg) | 1 | 3 | 0 | 4 | 2
  Decrease in systolic BP (>=30 mmHg) | 5 | 3 | 3 | 5 | 1
  Decrease in diastolic BP (>=20 mmHg) | 4 | 3 | 2 | 6 | 5

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 14 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to 14 days after last dose of study treatment (up to 101 days)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 61 | 60 | 61 | 61 | 61
participants
  AEs | 26 | 28 | 31 | 29 | 36
  SAEs | 0 | 1 | 2 | 1 | 1

8. Secondary Outcome: Percentage of Participants With at Least 1 Hypoglycemic Events (HAE) Episode
Description: A hypoglycemic event was identified by characteristic symptoms or blood glucose levels. HAE was defined as 1 of the given definitions: Characteristic symptoms of HAE with no home glucose monitoring performed where clinical picture included prompt resolution with food intake, subcutaneous glucagon, or intravenous glucose; or characteristic symptoms of HAE with home glucose monitoring measurement =< 70 milligram per deciliter (mg/dL) using ACCU-CHEK plasma-referenced home glucometers or =<74 mg/dL using International Federation of Clinical Chemistry (IFCC) referenced ACCU-CHEK or central laboratory glucometers; or any laboratory glucose value, meeting the following criterion with or without accompanying symptoms: =<49 mg/dL using ACCU-CHEK plasma-referenced home glucometers or =<53 mg/dL using IFCC referenced ACCU-CHEK or central laboratory glucometers.
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 61 | 60 | 61 | 61 | 61
percentage of participants | 4.9 | 3.3 | 4.9 | 6.6 | 34.4

9. Secondary Outcome: Number of Hypoglycemic Events (HAE) Episodes Per Participant
Description: A hypoglycemic event was identified by characteristic symptoms or blood glucose levels. Median of 1 and 2 events per participant was reported.
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: events per participant
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 61 | 60 | 61 | 61 | 61
events per participant | 0 [0 to 5] | 0 [0 to 2] | 0 [0 to 6] | 0 [0 to 9] | 0 [0 to 65]

10. Secondary Outcome: Time to Each Recurrent Hypoglycemic Events (HAE) Episode Per Participant
Description: Median recurrence time was not to be calculated when less than 50% of the participants in a given arm experienced 1 or more HAEs.
Time Frame: Baseline (Day 1) up to Week 14
Population: Data was not collected since this outcome measure was not analyzed due to infrequency of the occurrence of HAEs among the participants.
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Body Weight at Week 2, 4, 6, 8, 12 and 14
Time Frame: Baseline (Day 1), Week 2, 4, 6, 8, 12, 14 (follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure and 'n' signifies participants evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 59 | 57 | 58 | 61 | 60
kilogram (kg)
  Baseline (n=59, 57, 58, 61, 60) | 89.859 (21.9513) | 89.518 (20.5752) | 89.860 (21.4376) | 87.530 (19.2248) | 90.388 (17.9358)
  Change at Week 2 (n=59, 57, 58, 61, 58) | -0.402 (1.0127) | -0.069 (1.1309) | -0.028 (1.0557) | -0.021 (0.9504) | -0.024 (1.1295)
  Change at Week 4 (n=58, 56, 55, 59, 60) | -0.620 (1.2025) | -0.378 (1.2415) | -0.074 (1.2356) | -0.284 (1.2856) | 0.310 (1.3831)
  Change at Week 6 (n=57, 54, 55, 59, 56) | -0.564 (1.3880) | -0.604 (1.3153) | -0.228 (1.6697) | -0.290 (1.2669) | 0.473 (1.4922)
  Change at Week 8 (n=58, 54, 53, 58, 56) | -1.082 (1.7217) | -0.522 (1.5396) | -0.311 (2.2260) | -0.397 (1.1285) | 0.493 (1.7023)
  Change at Week 12 (n=56, 52, 53, 55, 54) | -1.529 (2.0906) | -0.685 (1.7244) | -0.961 (2.6114) | -0.545 (1.4004) | 1.211 (1.8771)
  Change at Week 14 (n=55, 51, 53, 55, 53) | -1.478 (2.0389) | -0.472 (2.0387) | -0.978 (2.7040) | -0.573 (1.6589) | 1.234 (1.7481)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 10 mg; Week 2: Treatment difference and 80 percent(%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, duration of type 2 diabetes mellitus (T2DM), time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.0898, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.33, 80% CI 2-sided [0.08 to 0.59], Standard Error of Mean 0.196
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0555, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.37, 80% CI 2-sided [0.12 to 0.62], Standard Error of Mean 0.195
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0585, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.37, 80% CI 2-sided [0.12 to 0.61], Standard Error of Mean 0.193
Statistical Analysis 4: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0454, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.39, 80% CI 2-sided [0.14 to 0.64], Standard Error of Mean 0.194
Statistical Analysis 5: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2819, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.25, 80% CI 2-sided [-0.05 to 0.55], Standard Error of Mean 0.235
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0319, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.51, 80% CI 2-sided [0.20 to 0.81], Standard Error of Mean 0.235
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1835, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.31, 80% CI 2-sided [0.01 to 0.60], Standard Error of Mean 0.231
Statistical Analysis 8: Comparison: Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.93, 80% CI 2-sided [0.63 to 1.22], Standard Error of Mean 0.231
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.9689, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = -0.01, 80% CI 2-sided [-0.35 to 0.33], Standard Error of Mean 0.266
Statistical Analysis 10: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.2221, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.32, 80% CI 2-sided [-0.02 to 0.67], Standard Error of Mean 0.265
Statistical Analysis 11: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.2774, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.28, 80% CI 2-sided [-0.05 to 0.62], Standard Error of Mean 0.261
Statistical Analysis 12: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 1.09, 80% CI 2-sided [0.76 to 1.43], Standard Error of Mean 0.263
Statistical Analysis 13: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0667, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.58, 80% CI 2-sided [0.17 to 0.98], Standard Error of Mean 0.314
Statistical Analysis 14: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0133, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.78, 80% CI 2-sided [0.38 to 1.19], Standard Error of Mean 0.314
Statistical Analysis 15: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0260, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.69, 80% CI 2-sided [0.29 to 1.08], Standard Error of Mean 0.308
Statistical Analysis 16: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 1.63, 80% CI 2-sided [1.23 to 2.02], Standard Error of Mean 0.310
Statistical Analysis 17: Comparison: Placebo vs PF-04937319 10 mg; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.0335, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.80, 80% CI 2-sided [0.32 to 1.28], Standard Error of Mean 0.374
Statistical Analysis 18: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.1557, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.53, 80% CI 2-sided [0.05 to 1.01], Standard Error of Mean 0.373
Statistical Analysis 19: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.0132, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.92, 80% CI 2-sided [0.45 to 1.39], Standard Error of Mean 0.368
Statistical Analysis 20: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 2.68, 80% CI 2-sided [2.20 to 3.15], Standard Error of Mean 0.370
Statistical Analysis 21: Comparison: Placebo vs PF-04937319 10 mg; Week 14 (Follow-up): Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, duration of T2DM, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.0158, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.96, 80% CI 2-sided [0.45 to 1.46], Standard Error of Mean 0.394
Statistical Analysis 22: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 11, analysis 21]; Test type: Superiority or Other; p = 0.2132, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.49, 80% CI 2-sided [-0.01 to 0.99], Standard Error of Mean 0.392
Statistical Analysis 23: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 11, analysis 21]; Test type: Superiority or Other; p = 0.0263, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.86, 80% CI 2-sided [0.37 to 1.36], Standard Error of Mean 0.387
Statistical Analysis 24: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 11, analysis 21]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 2.62, 80% CI 2-sided [2.12 to 3.12], Standard Error of Mean 0.390

12. Secondary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Hemoglobin,hematocrit,red blood cells(RBC) count:less than [<]0.8*lower limit of normal [LLN],platelets:<0.5*LLN/greater than [>]1.75*upper limit of normal [ULN],white blood cells(WBC):<0.6*LLN or >1.5*ULN,lymphocytes,total neutrophils:<0.8*LLN or >1.2*ULN, basophils,eosinophil,monocytes:>1.2*ULN;aspartate aminotransferase,alanine aminotransferase, alkaline phosphatase:>0.3*ULN,total protein,albumin:<0.8*LLN or >1.2*ULN;total bilirubin,direct bilirubin,indirect bilirubin:>1.5*ULN;triglycerides,cholesterol:>1.3*ULN, HDL:<0.8*LLN, LDL:>1.2*ULN,blood urea nitrogen,creatinine:>1.3*ULN,uric acid:>1.2*ULN;sodium: <0.95*LLN or >1.05*ULN,potassium,chloride,calcium,bicarbonate:<0.9*LLN or >1.1*ULN;creatine kinase:>2.0*ULN;glucose:<0.6*LLN or >1.5*ULN,urine WBC and RBC:>= 20/High Power Field [HPF]),urine epithelial cells (>=1 HPF),urine bacteria >20 high-powered field;qualitative urine glucose,urine blood to Hgb ratio (>=1);urine(protein,nitrite,mucus,leukocyte >=1 in urine dipstick test).
Time Frame: Baseline (Day 1) up to Week 14
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Number analyzed (Participants) | 60 | 60 | 60 | 61 | 61
participants | 56 | 52 | 56 | 54 | 51

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and nonserious in another subject, or 1 subject may have experienced both serious and nonserious event during study. AEs were also collected during the course of run-in period (metformin background therapy).
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 10 mg | PF-04937319 50 mg | PF-04937319 100 mg | Glimepiride
Serious Adverse Events (participants affected / at risk) | 4/361 | 0/61 | 1/60 | 2/61 | 1/61 | 1/61
Other Adverse Events (participants affected / at risk) | 63/361 | 26/61 | 28/60 | 31/61 | 29/61 | 36/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 500 mg (N=361) | Placebo (N=61) | PF-04937319 10 mg (N=60) | PF-04937319 50 mg (N=61) | PF-04937319 100 mg (N=61) | Glimepiride (N=61)
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 500 mg (N=361) | Placebo (N=61) | PF-04937319 10 mg (N=60) | PF-04937319 50 mg (N=61) | PF-04937319 100 mg (N=61) | Glimepiride (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 1 | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation decreased (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 4 | 2 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1 | 1 | 1
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 3 | 2 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 3 | 0 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 1 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 3 | 5 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypolipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 1 | 2 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Radicular pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 1
Balanitis (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 2 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.